CLINICAL TRIAL: NCT02229370
Title: Extracranial Carotid Artery Aneurysm Registry
Brief Title: Carotid Aneurysm Registry
Acronym: CAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: UMC Utrecht (Other)
Responsible Party: Principal Investigator, Gert Jan de Borst, MD PhD, UMC Utrecht
Other Study IDs: CAR2014
Record Dates: First submitted 2014-08-26; First posted 2014-09-01 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Extracranial Carotid Artery Aneurysm
Keywords: extracranial; carotid; artery; aneurysm; registry; CAR
MeSH Terms: conditions — Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — blood withdrawel
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ECAA: all patients diagnosed with an extracranial carotid artery aneurysm

SUMMARY:
To prospectively collect data on ECAA we designed the Carotid Aneurysm Registry (CAR). The aim of this study is to collect data on ECAA and its treatment to assess the natural history of ECAA and the success and safety of different treatment strategies.

DETAILED DESCRIPTION:
CAR is a prospective observational study, initiated by the Department of Vascular Surgery at University Medical Centre Utrecht (UMCU), The Netherlands. The study is descriptive in nature. The registry will be conducted according to the principles of the Declaration of Helsinki (64th WMA General Assembly, Fortaleza, Brazil, October 2013). The medical ethics committee of the UMCU has approved the study and all patients must give written informed consent before enrollment. Study enrolment is open to any patient diagnosed with an ECAA and ongoing.

Enrollment criteria: Participation in the CAR is intended for all subjects diagnosed with an ECAA irrespective of chosen treatment. Aneurysms are defined as 150% dilatation of the normal vessel diameter, or any saccular aneurysm. To be included, aneurysms must be located in the CCA, the external carotid artery or in the extracranial part of the ICA.To be included in the registry, patients need to be 18 years old. There are no additional exclusion criteria.

Intervention and follow-up:CAR does not interfere with the physician's treatment decision. Follow-up visits and imaging studies are scheduled as usual in their clinical practice, as this study does also not interfere with or influence the follow-up regimen.

Study endpoints:The primary endpoint of the CAR is freedom from aneurysm related symptoms at 30 days and at mid- and longterm follow-up. The secondary endpoint comprises treatment safety.

Endpoint monitoring:An endpoint adjudication committee, consisting of clinical experts, is set up to harmonize and standardize endpoint assessment and to determine whether the endpoints meet described criteria. This committee will review important subjective endpoints reported by trial investigators. The members of this committee are blinded to the treatment regime.

Data collection and monitoring: Data collected will be recorded through a web-based case report form (CRF). Data will be collected at baseline, at the moment of intervention, at the 30-day (or first postoperative) visit and during the follow-up phase. Data will remain at the UMCU in a secure environment.

This registry is a multicenter study. Statistical analysis: Statistical analyses will be performed using SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* Individual has one or more aneurysms of the extracranial carotid artery. Defined as 150% dilatation of the normal vessel diameter, or any saccular aneurysm.
* Individual is ≥18 years of age.
* Individual has signed informed consent

Exclusion Criteria:

* none

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participation in the CAR is intended for all subjects diagnosed with an extracranial carotid artery aneurysm irrespective of chosen treatment.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2014-06; Primary Completion 2019-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
aneurysms related symptoms | 5 years
  Aneurysm related symptoms such as ipsilateral stroke, TIA or compression. Disability is assessed by the Rankin scale.

SECONDARY OUTCOMES:
number of peri- and postoperative complications. | 30 days
  Treatment safety includes peri- and postoperative complications and registration of reinterventions performed within 30days after initial treatment. Complications include peripheral nerve dysfunction, local hematoma or infection, local pain or headache, TIA, stroke, local bleeding or aneurysm rupture and all-cause mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Gert Jan de Borst, MD, PhD, Principal Investigator — UMC Utrecht
Locations (1):
- University Medical Center Utrecht, Utrecht, Utrecht, Netherlands

REFERENCES:
- [Background] Welleweerd JC, Bots ML, Kappelle LJ, Rinkel GJ, Ruigrok YM, Baas AF, van der Worp HB, Vergouwen MD, Bleys RL, Hendrikse J, Lo TR, Moll FL, de Borst GJ. Rationale and design of the extracranial Carotid artery Aneurysm Registry (CAR). J Cardiovasc Surg (Torino). 2018 Oct;59(5):692-698. doi: 10.23736/S0021-9509.16.08637-7. Epub 2015 Feb 6. PMID 25658976
- [Background] Welleweerd JC, de Borst GJ; Carotid Aneurysm Registry Project Group. Extracranial carotid artery aneurysm: optimal treatment approach. Eur J Vasc Endovasc Surg. 2015 Mar;49(3):235-6. doi: 10.1016/j.ejvs.2014.11.007. Epub 2014 Dec 9. No abstract available. PMID 25500055
- [Background] Welleweerd JC, Nelissen BG, Koole D, de Vries JP, Moll FL, Pasterkamp G, Vink A, de Borst GJ. Histological analysis of extracranial carotid artery aneurysms. PLoS One. 2015 Jan 30;10(1):e0117915. doi: 10.1371/journal.pone.0117915. eCollection 2015. PMID 25635813
- [Background] Welleweerd JC, de Borst GJ, de Groot D, van Herwaarden JA, Lo RT, Moll FL. Bare metal stents for treatment of extracranial internal carotid artery aneurysms: long-term results. J Endovasc Ther. 2015 Feb;22(1):130-4. doi: 10.1177/1526602814566405. PMID 25775693
- [Background] Welleweerd JC, Moll FL, de Borst GJ. Technical options for the treatment of extracranial carotid aneurysms. Expert Rev Cardiovasc Ther. 2012 Jul;10(7):925-31. doi: 10.1586/erc.12.61. PMID 22908925
- See also: Click here for more information about this study: Carotid Aneurysm Registry — http://carotidaneurysmregistry.com